CLINICAL TRIAL: NCT05578092
Title: A Phase 1/2 Multiple Expansion Cohort Trial of the SOS1 Inhibitor MRTX0902 in Patients With Advanced Solid Tumors Harboring Mutations in the KRAS MAPK Pathway
Brief Title: A Phase 1/2 Study of MRTX0902 in Solid Tumors With Mutations in the KRAS MAPK Pathway
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA247-0004; CA247-0004 (Other: Bristol-Myers Squibb Protocol ID); 0902-001 (Other: Mirati Therapeutics Protocol ID)
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor; Advanced Solid Tumor; Non Small Cell Lung Cancer; Colo-rectal Cancer
Keywords: Non Small Cell Lung Cancer; NSCLC; Colorectal Cancer; CRC; EGFR; KRAS; SOS1; Solid Tumor; Advanced Solid Tumor; Malignant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colonic Neoplasms; Colorectal Neoplasms | interventions — adagrasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1/1B Monotherapy (Experimental): Dose Escalation/Evaluation
  Interventions: Drug: MRTX0902
- Phase 1/1B Combination Therapy (Experimental): Dose Escalation/Evaluation and Food Effect Assessment
  Interventions: Drug: MRTX0902; Drug: MRTX849
- Phase 2 (Experimental): MRTX0902 and adagrasib combination RP2D administered to separate cohorts of patients with selected solid tumor malignancies with KRAS G12C mutation to include the following: NSCLC, CRC, Other Solid Tumors
  Interventions: Drug: MRTX0902; Drug: MRTX849

INTERVENTIONS:
Drug: MRTX0902 — SOS1 inhibitor
Drug: MRTX849 — KRAS G12C inhibitor
  Other Names: adagrasib (KRAZATI)
  Arms: Phase 1/1B Combination Therapy; Phase 2

SUMMARY:
This is a Phase 1/2, open-label, multicenter, study evaluating the safety, tolerability, PK, PD, and anti-tumor activity of MRTX0902 alone and in combination with MRTX849 (adagrasib) in patients with advanced solid tumor malignancy harboring mutations in the KRAS-MAPK pathways.

DETAILED DESCRIPTION:
This first-in-human clinical trial will begin with an exploration of MRTX0902 dose and regimen. Once safety experience and PK data are available for the monotherapy regimen, dose escalation of the combination of MRTX0902 and adagrasib will be initiated, and will include a separate preliminary food effect assessments on MRTX0902 PK in combination with adagrasib. As potentially viable regimens are identified, Phase 1b expansion cohorts may be implemented to ensure collection of sufficient safety and PK information, and early evidence of clinical activity are available to recommend Phase 2 regimens. In Phase 2, separate cohorts of patients by histological diagnosis and/or baseline characteristics will be evaluated for the clinical activity and efficacy of MRTX0902 in combination with adagrasib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of a solid tumor malignancy with any of the following oncogenic mutations detected in tumor tissue or ctDNA by a sponsor-approved test:

  1. MRTX0902 monotherapy: known KRAS mutations, known annotated recurrent activating SOS1, PTPN11, class III BRAF, or EGFR mutation, or known annotated recurrent inactivating NF1 mutation;
  2. MRTX0902 and adagrasib combination therapy: KRAS G12C mutation.
* Unresectable or metastatic disease
* No available treatment with curative intent; standard treatment is not available or patient declines
* Presence of tumor lesions to be evaluated per RECIST 1.1:

  1. Phase 1 dose escalation, RECIST 1.1 measurable or evaluable disease
  2. Phase 1b and Phase 2 cohorts, RECIST 1.1 measurable disease
* Presence of a tumor lesion amenable to mandatory biopsy for pharmacodynamic evaluation at baseline and on-study unless Sponsor-confirmed as medically unsafe or infeasible.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate organ function

Exclusion Criteria:

* Active brain metastases or carcinomatous meningitis
* Prior treatment with a KRAS G12C inhibitor (for Phase 1b expansion for MRTX0902 and adagrasib combination, and Phase 2 cohorts only)
* History of significant hemoptysis or hemorrhage within 4 weeks of the first dose of study treatment.
* Major surgery within 4 weeks of first dose of study treatment
* History of pneumonitis or interstitial lung disease
* Ongoing need for medication with following characteristics: substrate of CYP3A; strong inducer or inhibitor or CYP3A and/or P-gp; strong inhibitors of BRCP and proton pump inhibitors
* Cardiac abnormalities
* History of intestinal disease, inflammatory bowel disease, major gastric surgery, or other gastrointestinal conditions (eg, uncontrolled nausea, vomiting, malabsorption syndrome) likely to alter absorption of study treatment or result in inability to swallow oral medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of Patients who Experience Dose-Limiting Toxicity | 21 Days
Phase1/1B: Number of patients who experience a treatment-related adverse event | Up to 2 years
Phase 2: Objective response rate (ORR) | 2 years
Phase 2: Duration of response (DOR) | 2 years
Phase 2: Progression free survival (PFS) | 2 years
Phase 2: Overall survival (OS) | 2 years

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve | Up to 4 days
  AUC - MRTX0902 and adagrasib
Time to achieve maximal plasma concentration | Up to 4 days
  Tmax - MRTX0902 and adagrasib
Maximum observed plasma concentration | Up to 4 days
  Cmax - MRTX0902 and adagrasib
Terminal elimination half-life | Up to 4 days
  t1/2 - MRTX0902
Apparent total plasma clearance when dosed orally | Up to 4 days
  CL/F - MRTX0902
Apparent volume of distribution when dosed orally | Up to 4 days
  Vz/F - MRTX0902

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (18):
- United States (17):
  - Local Institution - 001-108, New Haven, Connecticut
  - Local Institution - 001-119, Newark, Delaware
  - Local Institution - 001-111, Orlando, Florida
  - Local Institution - 001-103, Baltimore, Maryland
  - Local Institution - 001-110, Rochester, Minnesota
  - Local Institution - 001-115, Hackensack, New Jersey
  - Local Institution - 001-106, Cincinnati, Ohio
  - Local Institution - 001-109, Portland, Oregon
  - Local Institution - 001-116, Pittsburgh, Pennsylvania
  - Local Institution - 001-101, Nashville, Tennessee
  - Local Institution - 001-102, Nashville, Tennessee
  - Local Institution - 001-112, Dallas, Texas
  - Local Institution - 001-122, Fort Worth, Texas
  - Local Institution - 001-107, Houston, Texas
  - Local Institution - 001-123, Tyler, Texas
  - Local Institution - 001-104, Fairfax, Virginia
  - Local Institution - 001-105, Seattle, Washington
- Local Institution - 001-114, Rio Piedras, Puerto Rico

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT05578092.html